CLINICAL TRIAL: NCT02773147
Title: Effect of Vitamin B Substitution on Plasma NFL and Neurocognitive Performance in HIV-infected Individuals With Increased Plasma Homocysteine
Brief Title: Effect of Vitamin B on Plasma Neurofilament Light Protein (NFL) in HIV-infected Individuals With Increased Plasma Homocysteine
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-004311-20
Record Dates: First submitted 2016-05-12; First posted 2016-05-16 (Estimated); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: HIV
MeSH Terms: interventions — Vitamin B 12; Folic Acid; Pyridoxine

ARMS (2):
- Triobe (Experimental): Cyanocobalamin 0,5 mg. Daily for 24 months. Folate 0,8 mg. Daily for 24 months. Pyridoxine 3,0 mg. Daily for 24 months.
  Interventions: Drug: Cyanocobalamin; Drug: Folate; Drug: Pyridoxine
- Control (No Intervention)

INTERVENTIONS:
Drug: Cyanocobalamin
  Arms: Triobe
Drug: Folate
  Arms: Triobe
Drug: Pyridoxine
  Arms: Triobe

SUMMARY:
The purpose of this study is to investigate if B vitamin substitution have effect on NFL (neurofilament light protein) plasma levels and neurocognitive performance in HIV-infected individuals with increased plasma homocysteine

ELIGIBILITY:
Inclusion Criteria:

1. The ability to understand and give informed consent to participate.
2. HIV-1 infected with stable ART > 12 months
3. Plasma HIV-RNA < 50 copies/ml
4. Plasma homocysteine ≥ 12 μmol/L (subjects with < 12 μmol/L will be included in the analysis of secondary endpoint 3 (see 5.4).
5. Male or female, age 18 or older.

Exclusion Criteria:

1. Treatment with trimethoprim-sulfamethoxazole or methotrexate
2. Ongoing B6, B12 or folate substitution
3. Antiepileptic treatment
4. Small bowel or ventricular resection
5. Disturbed absorption in small bowel (Mb Crohn, untreated coeliac disease)
6. Ongoing neurological disease or severe psychiatric disease
7. Any malignant tumor in the history.
8. Severe ongoing infection or opportunistic infection
9. AUDIT > 7 for men and > 5 for women
10. MADRS > 20
11. Significant B12 or folate deficiency that indicate substitution (all subjects will be offered adequate substitution, they will be included in the analysis of secondary endpoint 3 (see 5.4)).
12. Pregnancy at screening visit, or planning pregnancy during study period is an exclusion criteria. (Not due to toxicity of Triobe, but to elevated risk of being prescribed B-vitamins outside of trial. If study object gets pregnant during study, she can continue the study but must be excluded if she starts treatment with other B-vitamin treatment than Triobe.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Declining NFL or decreased rate of increase of NFL | One year

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Gisslén, MD, PhD, Principal Investigator — Göteborg University
Locations (1):
- Department of Infectious Diseases, Sahlgrenska university hospital, Gothenburg, Sweden